CLINICAL TRIAL: NCT01218815
Title: Complete Infarct Related Artery Revascularization in Acute Myocardial Infarction Patients - CORAMI Trial
Brief Title: Complete Infarct Related Artery Revascularization
Acronym: CORAMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to very low enrollment rate the study was terminated.
Sponsor: Fundacja Ośrodek Badań Medycznych (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3.0/2010
Record Dates: First submitted 2010-10-01; First posted 2010-10-11 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Culprit lesion IRA Revascularization (Experimental): Primary PCI of culprit lesion in IRA with drug eluting stent (DES) and PCI of the other critical lesion in IRA with another DES
  Interventions: Procedure: IRA stenting in culprit lesion only
- Complete IRA revascularization (Active Comparator): Primary PCI of culprit lesion in IRA with DES stent
  Interventions: Procedure: IRA stenting

INTERVENTIONS:
Procedure: IRA stenting in culprit lesion only — stenting
  Arms: Culprit lesion IRA Revascularization
Procedure: IRA stenting — Complete IRA revascularization
  Arms: Complete IRA revascularization

SUMMARY:
CORAMI trial is a prospective, international, multicenter randomized study which will be performed in experienced invasive facility centres with 24/7 PCI (percutaneous coronary intervention) duty and patient enrollment will continue for 18 months (October 2010 - March 2012).The aim of the study is to compare strategy of complete vs target lesion-only primary PCI in IRA (infarct related artery) in STEMI (ST elevation myocardial infarction) patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of STEMI (according to ESC 2007 definition)
* Chest pain onset <12 hours
* signed informed consent
* Presence of two critical lesions requiring PCI in IRA (LAD - left anterior descending, Cx - circumflex, RCA - right coronary artery)
* Target/culprit lesion which requires immediate stenting (>50 - 100%) and second critical lesion (70-90%) with TIMI 3 flow after PCI of the 1st target/culprit lesion
* Over 18 years of age
* IRA diameter ≥ 2.5 mm

Exclusion Criteria:

* Terminal illness with life expectancy less <1 year or active cancer disease - Pregnancy or possibility of pregnancy
* Second critical lesion in IRA >90% or occlusion
* Contraindications to PCI or/and stent implantation
* Contraindications to DES stent implantation
* Lesion diameters unsuitable for intended stent platform
* Active bleeding or coagulopathy
* Patient in cardiogenic shock (<90mmHg SBP and/or requiring IABP - intraaortic balloon pump - or vasopressors) - Killip 4 class
* Patient has Left Bundle Branch Block (LBBB) or pacemaker rhythm
* No future patient cooperation expected
* Patient is participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
ST resolution in ECG (electrocardiogram) and MBG (myocardial blush grade) | in-hospital directly after PCI
  This is a combined end-point of ST - segment resolution >70% assessed directly after PCI
  + MBG 3 assessed directly after PCI (assessments by ECG and QCA Corelab).

SECONDARY OUTCOMES:
Clinical major ischemic events | 12-months
  1. Death at 12-month clinical follow-up
  2. Stent thrombosis at 12-month follow-up according to ARC definition
  3. reMI at 12 months
  4. urgent TVR at 12 months
Adverse events and complications during hospital stay | during patient index hospitalization (up to 7 days)
  1. Immediate in-hospital angiographic complications (at least one or more of the following: distal embolisation, no-reflow, slow-flow, acute coronary artery occlusion,artery perforation, tamponade, dissection type B and above)
  2. urgent in-hospital Target Vessel Revascularization (PCI and/or CABG - coronary artery bypass graft)

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Dudek, MD, PhD, Principal Investigator — Department of Interventional Cardiology, Jagiellonian University Medical College in Krakow, Poland
Locations (10):
- Poland (9):
  - I Katedra i Klinika Kardiologii, Warszawski Uniwersytet Medyczny, Warsaw, Banacha 1a
  - Krakowskie centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii, Carint Scanmed Sp. z o.o., Krakow, Kraków
  - Podkarpackie Centrum Interwencji Sercowo -Naczyniowych NZOZ, Sanok, Podkarpackie Voivodeship
  - SP ZZOZ Powiatowy Szpital Specjalistyczny, Stalowa Wola, Stalowa Wola
  - Pracownia Hemodynamiki Szpital im. E. Szczeklika, Tarnów, Szpitalna 13
  - Centrum Kardiologii Inwazyjnej GVM Carint, Ostrowiec Świętokrzyski, Szymanowskiego 11
  - Instytut Kardiologii im. Prymasa Tysiąclecia Stefana Kardynała Wyszyńskiego, Warsaw, Warszawa
  - Centrum Kardiologii Inwazyjnej GVM Carint, Oświęcim, Wysokie Brzegi 4
  - Department of Interventional Cardiology, Jagiellonian University Medical College, Krakow
- Departament of Cardiology, University Hospital, Ljubljana, Ljubljana, Ljubljana, Slovenia